CLINICAL TRIAL: NCT02551796
Title: Comparison of Early Changes in Ocular Surface and Inflammatory Mediators Among Lenticule Extraction, Laser in Situ Keratomileusis and Femtosecond Laser-assisted Laser in Situ Keratomileusis
Brief Title: Early Changes Among FLEx, LASIK and FS-LASIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xingwu Zhong, MD PhD, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-001
Record Dates: First submitted 2015-09-13; First posted 2015-09-16 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Myopia; Astigmatism
Keywords: lenticule extraction; laser in situ keratomileusis; femtosecond laser-assisted laser in situ keratomileusis; tear; inflammatory mediators
MeSH Terms: conditions — Myopia; Astigmatism; Lacerations | interventions — Tobramycin; Dexamethasone; Tobramycin, Dexamethasone Drug Combination; methylacetylene; Levofloxacin; Hyaluronic Acid; Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- lenticule extraction (Experimental): The patients in this group chose to receive the lenticule extraction surgery.
  Interventions: Procedure: lenticule extraction
- laser in situ keratomileusis (Experimental): The patients in this group chose to receive the laser in situ keratomileusis surgery.
  Interventions: Procedure: laser in situ keratomileusis
- FS assisted laser in situ keratomileusis (Experimental): The patients in this group chose to receive the FS assisted laser in situ keratomileusis surgery.
  Interventions: Procedure: FS assisted laser in situ keratomileusis

INTERVENTIONS:
Procedure: lenticule extraction — Four femtosecond incisions will be created in succession: the posterior surface of the refractive lenticule (spiral in), the lenticule border, the anterior surface of the refractive lenticule (spiral out), and the corneal flap in the superior region. After the suction is released, the flap will be opened using a thin, blunt spatula and the free refractive lenticule will be subsequently grasped with a forceps and extracted, after which the flap will be repositioned carefully.
  Other Names: 0.3% tobramycin/dexamethasone (TobraDex, Alcon); 0.5% levofloxacin (Cravit, Santen); sodium hyaluronate (HYCOSAN,URSAPHARM Arzneimittel GmbH)
  Arms: lenticule extraction
Procedure: laser in situ keratomileusis — During LASIK surgery, the eye will be gently proptosed and a hinged corneal flap will be cut using a microkeratome. The flap will be lifted and the stromal bed will receive a 6 mm diameter and stroma ablation. Finally reposition the flap carefully.
  Other Names: 0.3% tobramycin/dexamethasone (TobraDex, Alcon); 0.5% levofloxacin (Cravit, Santen); sodium hyaluronate (HYCOSAN,URSAPHARM Arzneimittel GmbH)
  Arms: laser in situ keratomileusis
Procedure: FS assisted laser in situ keratomileusis — Track distance and spot distance will be 3.0 μm during flap creation and 1.5 μm during flap side-cutting. The flap diameter will be 8.0 mm, and flap thickness will be set to 105 μm. Side-cut angle and hinge angle will be 90°and 50° respectively. The flaps will be created by laser scanning in spirals from the periphery to the center of the pupil. An excimer laser system will be used in the subsequent ablation of thstromal bed with a 6.0 mm optical zone. Once the excimer. ablation is completed, the flap will be repositioned in a similar fashion as in routine LASIK.
  Other Names: 0.3% tobramycin/dexamethasone (TobraDex, Alcon); 0.5% levofloxacin (Cravit, Santen); sodium hyaluronate (HYCOSAN,URSAPHARM Arzneimittel GmbH)
  Arms: FS assisted laser in situ keratomileusis

SUMMARY:
To evaluate the short-term changes in ocular surface measures and tear inflammatory mediators after lenticule extraction (FLEx), laser in situ keratomileusis (LASIK) and femtosecond laser-assisted laser in situ keratomileusis (FS-LASIK) procedures.

DETAILED DESCRIPTION:
Laser in situ keratomileusis (LASIK) with a microkeratome has been accepted wildly in the past 20 years. Gradually, laser in situ keratomileusis with a femtosecond laser-created flap (FS-LASIK)has been a popular ophthalmic procedure for the correction of refractive error. This first all-in-one FS-laser system was designed to perform the refractive lenticule extraction (ReLEx) procedures, femtosecond lenticule extraction (FLEx).They have the same feature: corneal flap.

Ocular surface disruption during corneal refractive surgery is commonly considered to be closely related to the development of dry eye. Multiple etiologies contribute to this ocular surface disruption, including the flap creation and stromal ablation involved in previous refractive surgery techniques. Corneal nerve damage has been considered the main cause of dry eye, due to disrupted afferent sensory nerves, reduced blink reflex, and increased tear evaporation leading to tear film instability. In addition, postoperative inflammatory mediator fluctuations are also a key factor related to ocular surface damage. Extensive research has described the effects of cytokines, chemokines and growth factors in modulating corneal wound healing, cell migration, and apoptosis on the ocular surface after refractive surgery.

This prospective clinical study is going to analyze the short-term changes in ocular surface measures and tear inflammatory mediators after FLEx, LASIK and FS-LASIK procedures.

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 18 years(range from 18 year to 31 years); corneal thickness 500 μm with calculated residual stromal bed after treatment greater than 300 μm; preoperative spherical equivalent refraction between
* 2.00 diopter (D) and -6.50 D; preoperative cylindrical equivalent refraction between -0.25 D and -1.50 D; preoperative corneal curvature from 42.0 D to 46.0 D with a regular topographic pattern, verified with an Atlas topographer; monocular best corrected visual acuity of 20/20 or better and stable refractive error (less than 0.5 D change) for 24 months before surgery

Exclusion Criteria:

* systemic disease that contraindicated the surgery (such as diabetes, glaucoma and systemic collagen vascular disease); corneal abnormality or disease; a history of tear supplement usage or contact lens wear during the past year

Ages: 18 Years to 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
scale of Schirmer I test | up to 1month after surgery
scale of corneal fluorescein staining | up to 1month after surgery
scale of noninvasive tear breakup time | up to 1month after surgery
questionnaire of ocular surface disease index | up to 1month after surgery
scale of central corneal sensitivity | up to 1month after surgery
scale of tear meniscus height | up to 1month after surgery
concentration of Interleukin-1α | up to 1month after surgery
concentration of tumor necrosis factor-α | up to 1month after surgery
concentration of nerve growth factor | up to 1month after surgery
interferon-γ | up to 1month after surgery
concentration of transforming growth factor-β1 | up to 1month after surgery
concentration of matrix metalloproteinase-9 | up to 1month after surgery

SECONDARY OUTCOMES:
Correlation between Interleukin-1α and ocular surface disease index | up to 1month after surgery
Correlation between tumor necrosis factor-α and ocular surface disease index | up to 1month after surgery
Correlation between nerve growth factor and ocular surface disease index | up to 1month after surgery
Correlation between interferon-γ and ocular surface disease index | up to 1month after surgery
Correlation between transforming growth factor-β1 and ocular surface disease index | up to 1month after surgery
Correlation between matrix metalloproteinase-9 and ocular surface disease index | up to 1month after surgery
Correlation between Interleukin-1α and corneal fluorescein staining | up to 1month after surgery
Correlation between tumor necrosis factor-α and corneal fluorescein staining | up to 1month after surgery
Correlation between nerve growth factor and corneal fluorescein staining | up to 1month after surgery
Correlation between interferon-γ and corneal fluorescein staining | up to 1month after surgery
Correlation between transforming growth factor-β1 and corneal fluorescein staining | up to 1month after surgery
Correlation between matrix metalloproteinase-9 and corneal fluorescein staining | up to 1month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xingwu Zhong, Principal Investigator — Hainan Eye Hospital, Zhongshan Ophthalmic Center of Sun Yat-sen University
Locations (1):
- Hainan Eye Hospital, Zhongshan Ophthalmic Center of Sun Yat-sen University, Haikou, Hainan, China